CLINICAL TRIAL: NCT05238584
Title: A Multicenter, Prospective, Randomized Trial to Evaluate the Role of Total Versus Partial Omentectomy in the Treatment of Tis - T3 Gastric Cancer.
Brief Title: Total Versus Partial Omentectomy in the Treatment of Gastric Cancer
Acronym: TOPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Debrecen (Other)
Collaborators: National Institute of Oncology, Hungary (Other); University of Pecs (Other); Uzsoki Hospital (Other)
Responsible Party: Principal Investigator, Dezso Toth, Associate Professor, University of Debrecen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOPO
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Stomach Neoplasms; Interleukin; Stomach Cancer; Gastric Cancer; Digestive System Neoplasm
Keywords: gastric cancer; total omentectomy; partial omentectomy; stomach cancer; interleukin; immunological answer
MeSH Terms: conditions — Stomach Neoplasms; Digestive System Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Total omentectomy (No Intervention): Total or subtotal gastrectomy with D2 lymphadenectomy and total omentectomy.
- Partial omentectomy (Experimental): Total or subtotal gastrectomy with D2 lymphadenectomy and partial omentectomy.
  Interventions: Procedure: Partial omentectomy

INTERVENTIONS:
Procedure: Partial omentectomy — Partial omentectomy: with preservation of the greater omentum at >2 cm from the gastroepiploic arcade.
  Arms: Partial omentectomy

SUMMARY:
The main purpose of this study is to evaluate the role of the type of omentectomy (partial or total) in the treatment of Tis - T3 gastric cancer without serosal infiltration. The second purpose is to monitoring the blood levels of immunological factors (interleukins, T cell subtypes, etc.) pre-and postoperatively, depending on the type of omentectomy.

DETAILED DESCRIPTION:
Gastric cancer is the second common tumor type. In 2020, the incidence of gastric cancer was over one million and caused about 770 000 tumor-associated deaths worldwide. Although the improvement of the perioperative oncological therapy is unquestionable, the major point of the treatment is radical surgical intervention. Laparoscopic technic is widespread in the treatment of gastric cancer, too. For the oncological radicality total or subtotal gastrectomy with D2 omentectomy is necessary, but the opinions are divided about the role of the omentectomy. Total omentectomy in laparoscopic operations takes more time and increases the postoperative morbidity, blood loss, and opportunity of the anastomosis insufficiency, and the incidence of the omental metastases is just between 3,8 - 5%. Based on this, many international guidelines allow partial omentectomy in early gastric cancer. At the same time, in advanced gastric neoplasm, the place of the partial omentectomy is still unclear.

With this prospective, randomized, multicentric study we plan to compare the total and partial omentectomy in the surgery of Tis - T3 gastric cancer with the analysis of the postoperative morbidity and mortality and long-term survival factors.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-III., Karnofsky Performance Score (KPS) >60, Eastern Cooperative Oncology Group (ECOG) 0-1
* Tis-T3 gastric cancer without serosal infiltration and treated with the radical operation (R0; D2 lymphadenectomy, lymph nodes >16)
* clinical stadium: Tis-3; M0
* written informed consent provided
* good patient compliance
* no previous chemotherapy or irradiation

Exclusion Criteria:

* serosal infiltration and/or distant metastasis, omental infiltration, peritoneal carcinosis, positive abdominal cytological lavage
* organ transplantation and/or immunological disease and/or immunomodulation therapy
* another primary tumor
* decompensated chronic disease (for example: liver cirrhosis with ascites, kidney failure treated with hemodialysis, New York Heart Association (NYHA) IV. cardiac status, etc.)
* unsuccessful follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
3y Overall Surveillance | 3 years
  Duration from the operation to the date of death.
3y Disease Free Surveillance | 3 years
  Duration from the operation to the date of radiological or histological proven relapse.

SECONDARY OUTCOMES:
Postoperative Complications (Clavien - Dindo classification) and morbidity | 30 days
  Incidence of 30 days postoperative morbidity (Clavien - Dindo classification).
Postoperative immunological changes (Interleukin monitoring) | 30 days
  Compare the pre-and postoperative interleukin blood levels to monitoring the immunological answer after total or partial omentectomy.

OTHER OUTCOMES:
Patient Data | 1 week
  Patient age, sex, BMI, etc.
Surgical Data | 1 week
  Duration of the operation, type of the operation (laparoscopic or open), intraoperative blood loss, etc.
Histopathological Data | 1 month
  Type of the tumor, TNM stadium, positive resection border, etc.
Duration of the hospital stay | 1 month
  The time from the date of operation to the date of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Dezső Tóth, Study Chair — University of Debrecen - Surgical Clinic
Locations (1):
- University of Debrecen - Surgical Clinic, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamabe A, Omori T, Tanaka K, Nishida T. Comparison of long-term results between laparoscopy-assisted gastrectomy and open gastrectomy with D2 lymph node dissection for advanced gastric cancer. Surg Endosc. 2012 Jun;26(6):1702-9. doi: 10.1007/s00464-011-2096-0. Epub 2011 Dec 30. PMID 22207307
- [Background] Zeng F, Chen L, Liao M, Chen B, Long J, Wu W, Deng G. Laparoscopic versus open gastrectomy for gastric cancer. World J Surg Oncol. 2020 Jan 27;18(1):20. doi: 10.1186/s12957-020-1795-1. PMID 31987046
- [Background] Ha TK, An JY, Youn HG, Noh JH, Sohn TS, Kim S. Omentum-preserving gastrectomy for early gastric cancer. World J Surg. 2008 Aug;32(8):1703-8. doi: 10.1007/s00268-008-9598-5. PMID 18536863
- [Background] Kim MC, Kim KH, Jung GJ, Rattner DW. Comparative study of complete and partial omentectomy in radical subtotal gastrectomy for early gastric cancer. Yonsei Med J. 2011 Nov;52(6):961-6. doi: 10.3349/ymj.2011.52.6.961. PMID 22028160
- [Background] Jongerius EJ, Boerma D, Seldenrijk KA, Meijer SL, Scheepers JJ, Smedts F, Lagarde SM, Balague Ponz O, van Berge Henegouwen MI, van Sandick JW, Gisbertz SS. Role of omentectomy as part of radical surgery for gastric cancer. Br J Surg. 2016 Oct;103(11):1497-503. doi: 10.1002/bjs.10149. Epub 2016 Aug 23. PMID 27550526
- [Background] Kim DJ, Lee JH, Kim W. A comparison of total versus partial omentectomy for advanced gastric cancer in laparoscopic gastrectomy. World J Surg Oncol. 2014 Mar 26;12:64. doi: 10.1186/1477-7819-12-64. PMID 24669875
- [Background] Japanese Gastric Cancer Association. Japanese gastric cancer treatment guidelines 2018 (5th edition). Gastric Cancer. 2021 Jan;24(1):1-21. doi: 10.1007/s10120-020-01042-y. Epub 2020 Feb 14. No abstract available. PMID 32060757
- See also: World Health Organisation (WHO) International Agency for Research on Cancer - Stomach — https://gco.iarc.fr/today/data/factsheets/cancers/7-Stomach-fact-sheet.pdf